CLINICAL TRIAL: NCT06202157
Title: Metabolic Differences Between Dihydroberberine and Micellar Berberine in Humans
Brief Title: Metabolic Differences Between Dihydroberberine and Micellar Berberine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Factors Group of Nutritional Companies Inc. (Industry)
Collaborators: Isura (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RR401
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Phase I and Phase II Metabolites of Berberine
Keywords: metabolites; berberine; micellar; dihydroberberine; pharmacokinetics
MeSH Terms: interventions — dihydroberberine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LMB (LipoMicel Berberine) (Experimental)
  Interventions: Other: LMB
- DHB (Dihydroberberine) (Experimental)
  Interventions: Other: DHB

INTERVENTIONS:
Other: LMB — A baseline blood sample (t=0) is collected from each participant prior to the intervention (LMB), and subsequent blood samples are collected at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours post-intervention.
  Other Names: LipoMicel Berberine
  Arms: LMB (LipoMicel Berberine)
Other: DHB — A baseline blood sample (t=0) is collected from each participant prior to the intervention (DHB), and subsequent blood samples are collected at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours post-intervention.
  Other Names: Dihydroberberine
  Arms: DHB (Dihydroberberine)

SUMMARY:
Differences in metabolites of dihydroberberine (DHB) and micellar berberine (LipoMicel®, LMB) are investigated through a randomized study involving human volunteers. Over a 24-hour period, blood samples are collected and subjected to Ultra High-Performance Liquid Chromatography-High Resolution Mass Spectrometry (UHPLC-HRMS) analysis to quantify the concentrations of berberine and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* healthy, good physical condition

Exclusion Criteria:

* Pregnancy or breast-feeding
* Gastrointestinal conditions
* Acute or chronic liver disease
* Acute or chronic kidney disease
* Acute or chronic cardiovascular disease
* Hematological disease
* Diabetes
* Allergy or Intolerance to gluten
* Allergy or Intolerance to Berberine
* Use of any form of nicotine or tobacco
* Alcohol and substance abuse history
* Use of medications (e.g., blood sugar-lowering agents, or statins)
* Use of Berberine supplements
* Participation in another investigational study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
AUC: the area under the concentration-time curve | at baseline (t=0 hours; before intervention), at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours post-intervention.
  For each berberine metabolite, PK parameters such as Area Under Curve (AUC) of the blood concentrations over a 24-hour period are reported.
Cmax: the maximum blood concentration | at baseline (t=0 hours; before intervention), at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours post-intervention.
  For each berberine metabolite, PK parameters such as the maximum blood concentration (Cmax) are reported.
Tmax: the time at which Cmax is reached | at baseline (t=0 hours; before intervention), at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours post-intervention.
  For each berberine metabolite, PK parameters such as Tmax, the time at which Cmax is reached, are reported.

CONTACTS AND LOCATIONS:
Locations (1):
- ISURA, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No